CLINICAL TRIAL: NCT06863597
Title: A Multi-Center Randomized, Parallel-Group Study to Compare Knowledge Translation Between Different Media in Pregnant and Lactating Women
Brief Title: Breastfeeding Advices on OTC Medicines With the Internet: What is the Best Medium
Acronym: LACT-ED
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 9/2024; BM/26617-3/2024 (Other: Hungarian Medical Research Council)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Breastfeeding Education; Lactating Mother; Breastfeeding Mothers; Lactation; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Masking Description: Blinding is not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Video content (Experimental): Participating mothers watch a video on a specific topic.
  Interventions: Other: Video content
- Written content (Experimental): Participating mothers read a text about a specific topic.
  Interventions: Other: Written content
- Podcast content (Experimental): Participating mothers listen to a podcast on a specific topic.
  Interventions: Other: Podcast content
- Illustration (information leaflet) content (Experimental): Participating mothers view an illustration on a specific topic.
  Interventions: Other: Illustration (information leaflet) content

INTERVENTIONS:
Other: Video content — Video content produced by media professionals using expert opinions.
  Arms: Video content
Other: Written content — Written content produced by healthcare professionals with experience in health education.
  Arms: Written content
Other: Podcast content — Podcast content created by media experts based on expert opinions.
  Arms: Podcast content
Other: Illustration (information leaflet) content — Illustration-based content created by media experts using expert opinions.
  Arms: Illustration (information leaflet) content

SUMMARY:
Pharmacotherapy for lactating women in Hungary presents a unique challenge. While certain medications may pose risks to the infant or reduce breast milk production, the unnecessary avoidance of treatment can also be harmful. Despite this, no dedicated Hungarian website currently provides guidance on the safe use of over-the-counter (OTC) medications for breastfeeding mothers.

To address this gap, the aim is to develop a website that not only meets clinical standards but also presents essential information in a clear, accessible format that helps mothers understand and retain key details by choosing the best medium.

Our main question is: What is the most effective way to educate lactating women about OTC medication use through an online platform?

ELIGIBILITY:
Inclusion Criteria:

* Target population is adult (>18 years), 3rd trimester pregnant women; and breastfeeding women after childbirth (max. 7 days postpartum; 24:00), who intend to breastfeed.
* Participants have to have internet access with no regard to the type of internet connection.

Exclusion Criteria:

* A mother will not breastfeed, either because they cannot or do not want it.
* Anyone who do not want to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Knowledge translation | From enrollment in the first week, followed by an assessment after 6 months.
  Knowledge translation will be measured by the difference in test scores before and after the intervention. The tests will be developed through common consensus. Since topic-specific tests will be created individually for each topic, only their utility will be assessed in a pilot study, and validation is not planned.

SECONDARY OUTCOMES:
User-satisfaction | From enrollment in the first week, followed by an assessment after 6 months.
  Questionnaire about user-satisfaction.

OTHER OUTCOMES:
Participating mother-specific features | From enrollment in the first week, followed by an assessment after 6 months.
  The questionnaire addresses topics related to baseline education and other factors that may influence the results.

CONTACTS AND LOCATIONS:
Overall Officials: Dénes Kleiner, PhD, Principal Investigator — Semmelweis University, University Pharmacy Department of Pharmacy Administration